CLINICAL TRIAL: NCT03743480
Title: Early Palliative Care and Hematological Cancer Patients: a Phase II Study
Brief Title: Early Palliative Care and Hematological Cancer Patients
Acronym: EPC-EMA1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/0056350
Record Dates: First submitted 2018-11-05; First posted 2018-11-16 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Neoplasms
Keywords: palliative care; cancer; hematologic malignancies
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Masking Description: centralized randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention): Patients in this arm will receive standard hematological care and palliative care on demand
- early palliative care (Experimental): early palliative care: patients in this arm will receive integrated palliative care
  Interventions: Other: early palliative care

INTERVENTIONS:
Other: early palliative care — experimental arm. Patients in this arm will meet with the palliative care team soon after the decision on their last active treatment
  Arms: early palliative care

SUMMARY:
The aim of the study is to pilot and evaluate a new integration model between a Specialised Palliative Care (SPC) intervention and standard hematological care in an Italian hospital. This is a feasibility mix-methods study, where a sample of advanced hematological patients are randomised to receive integrated hematological care and a SPC intervention or standard hematological care throughout the course of the predictive last active treatment.

DETAILED DESCRIPTION:
The most recent World Health Organization (WHO) definition of palliative care advocates that palliative care principles "…should be applied as early as possible in the course of any chronic, ultimately fatal illness". The difference with the previous WHO vision was substantial, as the earlier definition recommended Palliative Care to patients not responsive to curative therapy, limiting its role to the last period of life.

Evidence about the effectiveness of an early integration of palliative care has begun to emerge in the last years, primarily for cancer patients. The results of experimental studies, showed the effectiveness of early integration of palliative in the management of advanced illness, in improving quality of life, reducing consumption of resources, and possibly increasing survival. These data were also confirmed in Italy.

Hematological advanced patients suffer from a very high symptoms burden, psychological, spiritual, social and physical symptoms. They are very similar to oncological advanced patients. Hematologic patients during the last 30 days of their life are more frequently admitted in Hospital setting, emergency departments and high care ward than oncological patients, they received more aggressive treatments and more chemotherapy or biologic active treatments than oncologic patients.

Looking to WHO's palliative care definition and hematologic patients' symptoms burden it's simple to imagine that an early access to palliative care service could be the answer, as it was for advanced oncologic patients. The rational of the new vision lied on the recognition that palliative care had the potential to improve quality of life of patients and their family members during the whole trajectory of an incurable disease, through an effective management of psychological and physical symptoms, appropriate relationships, effective communication and support in decision-making.

In addition, even if WHO definition is referred to incurable patients, recent experience on Palliative care and Hematology is also about potentially curative patients.

Nonetheless, access to palliative care in hematologic patients care results totally absent or confined in the last days of life.There is a resistance by hematologic specialists to address patients to a palliative care service because of the possible misunderstanding between active treatment and palliative care assistance, identified from many professionals as terminal care A call to a new model of integration between palliative care and hematologic service is strong; for some authors just from the beginning of an advanced disease and for other authors modelled on the different patients' needs.

The aim of the study is to pilot a new model of integration for advanced hematological cancer between hematology and palliative care. Eligible patients will be at their last active treatment (chemotherapy or immunotherapy) as decided by hematologists.

The primary aim is to evaluate the feasibility, acceptability and efficacy of this novel intervention.

The evaluation procedure will be evaluated for feasibility and applicability To the investigators knowledge this is the first trial on an integrative model between palliative care and hematology for an advanced hematological population.

Primary aim

To evaluate the feasibility of integrated versus standard involvement of palliative team for hematological advanced patients.

Secondary aims to evaluate the efficacy of this new model on Quality of Life (QoL) until 6 months after the enrollment.

to evaluate the impact of the intervention on care pathways (number of chemotherapies in the last 30 days, number of exams, length of stay in Hospital or Hospice, access to emergency department, setting of death and so on) to evaluate the acceptability of the intervention by patients, professionals and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed incurable hematological tumor;
* Estimated prognosis by the hematologist more than 1 month at least;
* Predictive last active treatment (chemotherapy or immunotherapy) as established by hematological team;
* 18 years old;
* Eastern Cooperative Oncology Group ≤ 3;
* Ability to read and respond to questions in Italian;
* Consent to the study

Exclusion Criteria:

* Existence of other co morbid disease which in the opinion of the investigator prohibits participation in the protocol;
* Caregiver's absence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Adherence to the palliative care program assessed by percentage of patients attending palliative care visits after 3 months from the enrolment | 3 months after the enrollment
  the investigators consecutively register all eligible patients (and reasons for ineligibility) both from Hematological department, patients who were asked to participate to the study (and reasons for not), patients who accepted to participate (and reasons for not). The feasibility will be achieved if >50% of patients remain in the program in the next 3 months from the enrollment

SECONDARY OUTCOMES:
Quality of life of patients assessed by Palliative Care Outcomes Scale | At the time of the randomization, after 4 weeks from the randomization and then every 4 weeks for 6 months
  The efficacy on QoL during the follows 6 months will be assessed by Palliative Care Outcomes Scale. range 0-40,higher value means worse outcome
quality of life of patients assessed by symptoms control 'measurement | At the time of the randomization, after 4 weeks from the randomization and then every 4 weeks for 6 months
  1. The efficacy on QoL during the follows 6 months will be assessed by Edmonton Symptom Assessment System. Range 0-100. Higher value means worse outcomes
incidence of anxiety and depression between patients enrolled | At the time of the randomization, after 4 weeks from the randomization and then every 4 weeks for 6 months
  assessed by
  - Hospital Anxiety and Depression Scale,range 0-42, higher value means worse outcomes
Performance status changing during the program | At the time of the randomization, after 4 weeks from the randomization and then every 4 weeks for 6 months
  during the follows 6 months will be assessed by Eastern Cooperative Oncology Group. It measures performance status, range 0-5, higher value worse outcomes
Qualitative evaluation by patients/caregivers on palliative care program | After 12 weeks from the randomization for patients or caregivers. Investigators establish as necessary that patients have attended 3 palliative care visits. Professionals will be interview at the end of the enrolment
  individual semi-structured interviews exploring the experience of the different 'actors' of the intervention, i.e. the receivers (patients and family members) and professionals. Semistructured interviews are in deep interviews and they are not linked to a scale

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Tanzi, MD, Principal Investigator — Azienda USL Reggio Emilia - IRCCS
Locations (2):
- Italy (2):
  - Arcispedale santa maria nuova-viale risorgimento 80, Reggio Emilia, Emilia-Romagna
  - Viale Risorgimento 80, Reggio Emilia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanzi S, Luminari S, Cavuto S, Turola E, Ghirotto L, Costantini M. Early palliative care versus standard care in haematologic cancer patients at their last active treatment: study protocol of a feasibility trial. BMC Palliat Care. 2020 Apr 22;19(1):53. doi: 10.1186/s12904-020-00561-w. PMID 32321483

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT03743480/Prot_SAP_000.pdf